CLINICAL TRIAL: NCT02979574
Title: Personalize Electro-acupuncture vs. Auricular-acupuncture Comparative Effectiveness
Brief Title: PEACE: Comparing Chronic Pain Treatment Options
Acronym: PEACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-1579
Record Dates: First submitted 2016-11-28; First posted 2016-12-01 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Musculoskeletal Pain; Fibromyalgia; Pain Management
Keywords: acupuncture; pain; chronic pain; pain management; 16-1579
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Fibromyalgia; Agnosia; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Electro-Acupuncture (EA) Procedure (Active Comparator): Participants will receive 10 treatment of EA acupuncture over the course of 10 weeks (with a maximum of 2 treatments per week).
  Interventions: Procedure: Electro-Acupuncture (EA)
- Battle Field Acupuncture (BFA) Procedure (Active Comparator): Participants will receive 10 treatment of BFA acupuncture over the course of 10 weeks (with a maximum of 2 treatments per week).
  Interventions: Procedure: Battle Field Acupuncture (BFA)
- Wait List Control (WLC) Usual Care Procedure (Active Comparator): Subjects in the WLC group continue to receive their standard medical care and pain management as prescribed by their physicians or other health care providers, including analgesic medications. After the 12 week follow up period, patients in the WLC will receive up to ten treatments of either EA or BFA based on their personal preference.
  Interventions: Procedure: Electro-Acupuncture (EA); Procedure: Battle Field Acupuncture (BFA); Device: Wait List Control (WLC)

INTERVENTIONS:
Procedure: Electro-Acupuncture (EA) — Participants will receive 10 treatment of Electro-Acupuncture over the course of 10 weeks (with a maximum of 2 treatments per week). The acupuncturist will insert acupuncture needles in at least 4 local points around the body with the most pain and at least 4 distant points to address the patient's baseline constitution. The needles will be electrically stimulate at 2 Hz by connecting to a TENS unit. The needles will be in place for 30 minutes.
  Arms: Electro-Acupuncture (EA) Procedure; Wait List Control (WLC) Usual Care Procedure
Procedure: Battle Field Acupuncture (BFA) — Participants will receive 10 treatment of Battle Field Acupuncture over the course of 10 weeks (with a maximum of 2 treatments per week). Acupuncture needles will be placed in the participants' ears. The total duration of BFA delivery is about 10 to 20 minutes depending on how many needles are used in the procedure.
  Arms: Battle Field Acupuncture (BFA) Procedure; Wait List Control (WLC) Usual Care Procedure
Device: Wait List Control (WLC) — After the waiting period (12 weeks from randomization), participants in the WLC will receive up to ten treatments of either EA or BFA based on their personal preference.
  Arms: Wait List Control (WLC) Usual Care Procedure

SUMMARY:
The purpose of this study is to compare two types of acupuncture with usual care on treating chronic pain. This study has three groups. Two groups will received acupuncture. One group will receive usual standard of care for 12 weeks and then will receive acupuncture. Acupuncture is an ancient Chinese technique of using very thin needles inserted in the skin to treat different symptoms and illness, and to promote healing. Each group will undergo a different method of needle administration.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Age >/= 18 years or older
* Having musculoskeletal pain, defined as regional (joints, extremities, back, neck) or more generalized (fibromyalgia or chronic widespread pain)
* Having a pain rating of 4 or greater in worst pain on a 1-10 numerical rating scale in the preceding week (Patients with a neuropathic component to their pain that involves the extremities or back will be eligible)
* Having had pain for at least 3 months and at least 15 days with pain in the preceding 30 days
* A diagnosis of cancer with no restrictions placed on type of cancer, other than that patients with metastatic disease will be excluded. Eligibility criteria are not restricted to MSK confirmed biopsy/diagnosis. Participating institution's testing is sufficient for other study sites.
* Complete active treatment (surgery, chemotherapy, and/or radiotherapy) at least one month prior to study initiation (patients on continued hormone treatment will not be excluded).

Exclusion Criteria:

* Have non-musculoskeletal pain syndromes (headache, facial pain, chest pain, visceral abdominal pain) if these are the sole source of pain, but can be present as co-morbid conditions as long as a patient has a primary musculoskeletal pain condition defined s above.
* Inflammatory arthritis that require disease modifying drugs (e.g. rheumatoid arthritis)
* Phantom limb pain
* Patients with a history of metastatic cancer who are not currently NED
* Have a pending pain-related VA or social security or worker's comp disability claim by self-report
* Have an implanted electronically charged medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and pain interference will be measured by using the Brief Pain Inventory (BPI) measure. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li X, Lampson K, Rosa WE, Li QS, Ramalingam MB, Epstein AS, Mao JJ. Effect of acupuncture on fatigue in cancer survivors with chronic pain: a secondary analysis. Support Care Cancer. 2025 Dec 13;34(1):31. doi: 10.1007/s00520-025-10219-z. PMID 41389238
- [Derived] Booher A, Mao JJ, Muniz RC, Romero SAD, Li SQ, Lopez AM, Liou KT. Association between Hispanic Ethnicity and Greater Expectation of Benefit from Acupuncture or Massage for Pain in Cancer. J Immigr Minor Health. 2024 Oct;26(5):953-957. doi: 10.1007/s10903-024-01611-8. Epub 2024 Jul 8. PMID 38977653
- [Derived] Bao T, Zhi WI, Baser RE, Li QS, Weitzman M, Gillespie EF, Robson M, Mao JJ. Electro-acupuncture versus battle field auricular acupuncture in breast cancer survivors with chronic musculoskeletal pain: subgroup analysis of a randomized clinical trial. Breast Cancer Res Treat. 2023 Nov;202(2):287-295. doi: 10.1007/s10549-023-07072-1. Epub 2023 Aug 24. PMID 37612534
- [Derived] Mao JJ, Liou KT, Baser RE, Bao T, Panageas KS, Romero SAD, Li QS, Gallagher RM, Kantoff PW. Effectiveness of Electroacupuncture or Auricular Acupuncture vs Usual Care for Chronic Musculoskeletal Pain Among Cancer Survivors: The PEACE Randomized Clinical Trial. JAMA Oncol. 2021 May 1;7(5):720-727. doi: 10.1001/jamaoncol.2021.0310. PMID 33734288
- [Derived] Liou KT, Baser R, Romero SAD, Green J, Li QS, Orlow I, Panageas KS, Mao JJ. Personalized electro-acupuncture versus auricular-acupuncture comparative effectiveness (PEACE): A protocol of a randomized controlled trial for chronic musculoskeletal pain in cancer survivors. Medicine (Baltimore). 2020 May 22;99(21):e20085. doi: 10.1097/MD.0000000000020085. PMID 32481275
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/